CLINICAL TRIAL: NCT01547273
Title: The Effect of Bone and Connective Tissue Grafts on Facial Gingival Profile in Single Maxillary Anterior Immediate Implant Placement and Provisionalization: A 1-Year Prospective Study
Brief Title: The Effect of Bone Grafts on Facial Gingival Profile in Maxillary Anterior Single Tooth Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: DentiumUSA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 5110339
Record Dates: First submitted 2012-01-12; First posted 2012-03-07 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Facial Gingival Profile

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bone graft inside socket only (Experimental): bone graft inside socket only
  Interventions: Procedure: bone graft inside socket only
- bone graft inside and outside socket (Experimental): bone graft inside and outside socket
  Interventions: Procedure: bone graft inside and outside socket
- no bone graft (Experimental): no bone graft
  Interventions: Procedure: no bone graft

INTERVENTIONS:
Procedure: bone graft inside socket only — bone graft inside socket only
  Arms: bone graft inside socket only
Procedure: bone graft inside and outside socket — bone graft inside and outside socket
  Arms: bone graft inside and outside socket
Procedure: no bone graft — no bone graft
  Arms: no bone graft

SUMMARY:
The purpose of this investigator-initiated study is to evaluate the facial gingival profile following immediate implant placement and provisionalization in conjunction with connective tissue graft with or without bone graft

DETAILED DESCRIPTION:
Thirty subjects who are at least 18 years old with a failing upper front tooth seeking for implant treatment will be recruited at Loma Linda University School of Dentistry (LLUSD), where the consent will also take place. The subjects will be randomly divided into 3 groups. The subjects will receive immediate implant placement and provisionalization (IIPP) in conjunction with connective tissue graft (CTG) with (Group I) or without (Group II) bone graft in the extraction socket; and with bone graft in extraction socket and at the facial aspect of failing tooth (Group III). Clinical, radiographic and model assessments will be performed at different time intervals (pre-treatment to 12 months after implant placement) and statistically analyzed (α = 0.05) to evaluate peri-implant tissue response and facial gingival profile of the implants. Complications, if any, will also be recorded and appropriately addressed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older, are no longer growing and able to read and sign an informed consent.
2. Good oral hygiene.
3. A single failing maxillary anterior tooth (#6-11) with the presence of healthy adjacent teeth.
4. Adequate bone volume to accommodate an implant with minimum dimensions of 3.6 mm diameter and 10.0 mm length.
5. Presence of opposing dentition (natural teeth, fixed or removable prostheses)
6. Healthy soft tissue at the future implant site.

Exclusion Criteria:

1. A medical history that would complicate the outcome of study such as alcohol or drug dependency, poor health ,uncontrolled diabetes, immunodeficiency diseases, taking any medication that may cause gingival over growth or any other medical, physical or psychological reason that might affect the surgical procedure or the subsequent prosthodontic treatment and required follow-up examinations.
2. Dental history of bruxism, parafunction habit, and/or lack of stable posterior occlusion
3. Smoker.
4. History of head and neck radiation.
5. Soft tissue defect (inflammation, tissue cleft, unhealthy tissue) around a future implant site.
6. Inability to achieve primary implant stability following immediate implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03-20 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2016-04-07 (Actual)

PRIMARY OUTCOMES:
change in facial gingival profile | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joseph YK Kan, DDS, MS, Principal Investigator — Loma Linda University School of Dentistry
Locations (2):
- United States (2):
  - Implant Department, School of dentistry, Loma Linda University, Loma Linda, California
  - Loma Linda University School of Dentistry, Loma Linda, California